CLINICAL TRIAL: NCT01646216
Title: Long Term Split Belt Treadmill Training for Stroke Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); University of Maryland (Other); VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy J. Bastian, Ph.D., Dr. Amy J Bastian, Ph.D., PT, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00068967; 2P30AG028747-06 (NIH)
Record Dates: First submitted 2012-04-05; First posted 2012-07-20 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Stroke; Hemiparesis
Keywords: stroke; treadmill; walking; hemiparesis; training
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: Split belt treadmill
Oversight: Data Monitoring Committee: No

ARMS (1):
- Split-belt treadmill training (Experimental): Split-belt treadmill exercise
  Interventions: Behavioral: Split belt treadmill

INTERVENTIONS:
Behavioral: Split belt treadmill — A split belt treadmill is like a typical treadmill that is seen in the gym, except that this treadmill has two belts that move instead of just one. One leg goes on one belt and the other leg uses the other belt. The belt speeds can be set to move at the same speed, making this treadmill similar to any regular treadmill, but, belt speeds can also be set so that one belt moves a little faster than the other. The belts are never set at a running or jogging speed, only a self-paced walking speed regardless of whether the belts are both going the same or slightly different speeds.
  Other Names: Woodway Split Belt Treadmill; Company: Woodway USA, Inc

SUMMARY:
The purpose of this study is to determine whether split belt or conventional treadmill training can be used to treat walking pattern deficits from stroke and to determine whether this improves gait asymmetry and metabolic efficiency.

DETAILED DESCRIPTION:
Coordination between the legs during walking is often disrupted after neurological injury, resulting in asymmetric gait patterns. Recent data shows that walking patterns can be altered through treadmill training, even after central nervous system damage. The investigators have studied short-term adaptation of inter-limb coordination during walking using a split-belt treadmill to control speed of the two legs independently. Our findings demonstrate that walking patterns are adaptable. The investigators have also shown that people with cerebral damage from stroke can benefit in the short-term to correct asymmetric walking patterns. Since all of our previous work has focused on single training sessions or up to 4 week training sessions, the investigators would like to study long-term effects of split belt treadmill training. Therefore, the purpose of this study is to prepare for a clinical trial of split-belt treadmill training to treat walking pattern deficits from cerebral damage. The investigators will gather data to determine whether different types of treadmill training on a custom split-belt treadmill are likely to change/improve walking symmetry as well as metabolic efficiency.

The investigators will study adults with cerebral damage due to stroke. Subjects with hemiparesis will undergo training 3 times a week for a total of 33 training session. These 33 sessions will be broken into 3 blocks of 11 sessions. After each block of 11 sessions an evaluation will be done to record any gait improvements. Training for the subjects with hemiparesis will either be conventional treadmill walking (both legs moving at the same speed) or split-belt treadmill walking (with one leg moving faster than the other). These studies will provide important new information about normal mechanisms of locomotor adaptation, as well as providing a new rehabilitation tool for people with asymmetric gait patterns. Note that this study is not an aerobic conditioning program since subjects will work well below their age-adjusted target heart rate; it is instead a retraining program aimed at teaching people a new inter-limb coordination pattern as well as to determine whether this training can influence the subject's body's ability to use its intake of oxygen more efficiently. This study is also critical for developing procedural reliability processes, calculating effect sizes, training clinical staff, and determining other salient clinical variables in preparation for a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* stroke or hemiparesis (>6 months post stroke)
* able to walk but has residual gait deficit (including those who walk with a cane or walker)
* This is their first and only stroke
* Able to walk for 5 minutes at their self-paced speed
* Adults age 20-80

Exclusion Criteria:

* Cerebellar signs (e.g.ataxic hemiparesis)
* Any neurologic condition other than stroke
* Insulin dependent diabetes
* Congestive heart failure
* Peripheral artery disease with claudication
* Pulmonary or renal failure
* Unstable angina
* Uncontrolled hypertension (>190/110 mmHg)
* Dementia
* Severe aphasia
* Orthopedic or pain conditions that limit walking
* Total joint replacement in the lower extremities
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-06-07 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Bastian, PhD, PT, Principal Investigator — Kennedy Krieger Institute and Johns Hopkins School of Medicine
Locations (1):
- Motion Analysis Lab in the Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- See also: Link Text: Motion Analysis Lab website at the Kennedy Krieger Institute — http://www.kennedykrieger.org/kki_research.jsp?pid=5741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects recruited were 6 months or more post stroke. During 2012-2016 recruitment was done by the following means: Subjects were referred by local physicians and recruited from databases of previous studies. Flyers were disseminated locally. Presentations were made at local stroke support groups.
Pre-assignment Details: Subjects were enrolled and randomly assigned to either Split or Tied treadmill training groups.
Groups:
- Split-belt Treadmill Exercise: Split-belt treadmill training
  Split belt treadmill: A split belt treadmill is like a typical treadmill that is seen in the gym, except that this treadmill has two belts that move instead of just one. One leg goes on one belt and the other leg uses the other belt. The belt speeds can be set to move at the same speed, making this treadmill similar to any regular treadmill, but, belt speeds can also be set so that one belt moves a little faster than the other. The belts are never set at a running or jogging speed, only a self-paced walking speed regardless of whether the belts are both going the same or slightly different speeds.
- Tied-belt Treadmill Exercise: Tied-belt treadmill training
  The treadmill is run like a typical treadmill that is seen in the gym except that this treadmill has two belts that move instead of just one. One leg goes on one belt and the other leg uses the other belt. The belt speeds are set to move at the same speed, making this treadmill training group similar to any regular treadmill.
Period: Overall Study
Arm/Group | Split-belt Treadmill Exercise | Tied-belt Treadmill Exercise
Started | 17 | 17
Completed | 6 | 4
Not Completed | 11 | 13
Not completed — Baseline step length difference (<5cm) | 10 | 10
Not completed — Did not complete training | 0 | 2
Not completed — Investigator decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Split-belt Treadmill Exercise | Tied-belt Treadmill Exercise | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (11.7) | 59.2 (14.3) | 60 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Step Length Symmetry. That is, Whether the Steps With Right and Left Legs Are the Same Length.
Description: Subjects will either walk on a special mat that records their step lengths, or will wear special markers on the feet and body to record their step lengths.
Time Frame: After training (week 14), and 3 months after training
Population: Subjects were grouped by baseline walking speed into three levels of disability: mild, moderate, and severe.
Measure: Mean (Full Range); unit: ratio
Groups:
- Split-belt, Mild Disability: Subjects trained on split belt treadmill. Subjects in the mild disability group had baseline walking speeds greater than 0.8 m/s. There were two subjects in this group.
- Split-belt, Moderate Disability: Subjects trained on split belt treadmill. Subjects in the moderate disability group had baseline walking speeds of 0.4 m/s to 0.8 m/s. There were two subjects in this group.
- Split-belt Severe Disability: Subjects trained on split belt treadmill. Subjects in the severe disability group had baseline walking speeds less than 0.4 m/s. There were two subjects in this group.
- Tied-belt, Severe Disability: Subjects trained on tied belt treadmill. Subjects in the severe disability group had baseline walking speeds less than 0.4 m/s. There were three subjects in this group.
- Tied-belt Mild Disability: Subjects trained on tied belt treadmill. Subjects in the mild disability group had baseline walking speeds greater than 0.8 m/s. There was one subject in this group.
Arm/Group | Split-belt, Mild Disability | Split-belt, Moderate Disability | Split-belt Severe Disability | Tied-belt, Severe Disability | Tied-belt Mild Disability
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 1
ratio
  Post training | 0.001 [0.001 to 0.001] | -0.078 [-0.101 to -0.055] | -0.045 [-0.057 to -0.033] | 0.144 [-0.765 to 0.233] | -0.034 [-0.034 to -0.034]
  Follow up | 0.010 [0.007 to 0.013] | -0.075 [-0.091 to -0.058] | -0.124 [-0.221 to -0.028] | -0.096 [-0.412 to 0.125] | -0.027 [-0.027 to -0.027]

2. Secondary Outcome: Change in Baseline Oxygen Intake
Description: This is the change in metabolic power that is required of a subject to walk at their self selected walking speed on the treadmill. Metabolic power was measured at baseline, post training, and three months after training. We report the difference between post training and baseline and three months and baseline.
Time Frame: Post training (week 14), and 3 months follow up
Population: One subject in the Split-belt Severe Disability" Arm/Group did not complete the assessment during the change at follow up visit. Two subjects in the Tied-belt, Severe Disability Arm/Group were not able to complete the assessments at post training or follow up.
Measure: Mean (Full Range); unit: ml/kg/min
Arm/Group | Split-belt, Mild Disability | Split-belt, Moderate Disability | Split-belt Severe Disability | Tied-belt, Severe Disability | Tied-belt Mild Disability
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 1
ml/kg/min
  Change at post training: number analyzed (Participants) | 2 | 2 | 2 | 1 | 1
  Change at post training | 0.82 [0.13 to 1.5] | -.61 [-.79 to -.43] | 0.65 [-.59 to 1.89] | 4.616 [NA to NA] — Two subjects were not able to complete this assessment. | -2.272 [NA to NA] — There is only one subject in this group.
  Change at follow up: number analyzed (Participants) | 2 | 2 | 1 | 1 | 1
  Change at follow up | 0.86 [0.26 to 1.46] | -0.84 [-0.9 to -0.79] | -0.85 [-0.85 to NA] — One subject was not able to complete this assessment. | 4.009 [NA to NA] — Two subjects were not able to complete this assessment. | -2.675 [NA to NA] — There is only one subject in this group.

3. Secondary Outcome: Walking Speed
Description: Subjects walked on an electronic walkway and walking speed was calculated by total distance divided by total time.
Time Frame: Baseline, post training, and 3 month follow up.
Population: All subjects for whom walk speed was recorded at baseline, post training, and follow up.
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Split-belt, Mild Disability | Split-belt, Moderate Disability | Split-belt Severe Disability | Tied-belt, Severe Disability | Tied-belt Mild Disability
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 1
meters per second (m/s)
  Baseline | 1.22 (0) | 0.5 (0.09) | 0.11 (0.02) | 0.12 (0.06) | 1.08 (0)
  Post training | 1.17 (0.02) | 0.55 (0.10) | 0.16 (0.01) | 0.18 (0.02) | 1.10 (0)
  Follow-up (3 months) | 1.15 (0.02) | 0.63 (0.26) | 0.15 (0.02) | 0.16 (0.05) | 1.22 (0)

ADVERSE EVENTS:
Time Frame: 4 years, 9 months
Arm/Group | Split-belt Treadmill Exercise | Tied-belt Treadmill Exercise
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

LIMITATIONS AND CAVEATS:
Some subjects could not complete all of the tasks. Recruitment was also challenging.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT01646216/Prot_SAP_000.pdf